CLINICAL TRIAL: NCT00739947
Title: A PROSPECTIVE STUDY TO EVALUATE SURGICAL OUTCOMES IN SUBJECTS WITH FULL-THICKNESS ROTATOR CUFF TEARS TREATED BY MEANS OF A DOUBLE-ROW ARTHROSCOPIC REPAIR.
Brief Title: Arthroscopic Surgical Outcome Study In Subjects With Rotator Cuff Tears
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 3202V1-1000; B1861001 (Other: Alias Study Number)
Record Dates: First submitted 2008-08-21; First posted 2008-08-22 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Rotator Cuff; Arthroscopic Surgery
Keywords: Observational; rotator cuff tear; arthroscopic; surgical; outcome study
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Standard of Care
  Interventions: Other: Observational study of the surgical outcome

INTERVENTIONS:
Other: Observational study of the surgical outcome — Subjects return for 7 follow-up visits following arthroscopic repair of their rotator cuff. During the follow-up visits subjects undergo imaging with MRI and ultrasound.

SUMMARY:
This is an observational study that involves subjects with full-thickness rotator cuff tears treated by means of arthroscopy surgical repair, also known as arthroscopic surgery. The primary objective of this study is to observe the timing and rate of tendon retear in those subjects.

DETAILED DESCRIPTION:
Subjects will be recruited from each surgeon's surgical practice. They will be reviewed to assure they meet all eligibility criteria prior to enrolling them into the study.

ELIGIBILITY:
Inclusion Criteria:

* Full thickness Rotator Cuff Tears ranging from 1cm to 4cm in size.
* Planned procedure for repair is tendon-to-bone repair by means of an arthroscopy

Exclusion Criteria:

* Previous surgical intervention to the shoulder joint understudy
* Tears of the subscapularis or labral pathology requiring surgical repair
* Shoulder instability either shoulder
* Unable to complete functional evaluations in either shoulder

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2008-10-13 (Actual); Primary Completion 2011-07-05 (Actual); Study Completion 2011-07-05 (Actual)

PRIMARY OUTCOMES:
The primary objective is to observe the rate and timing of tendon retear in subjects with full thickness rotator cuff tears (RCTs) treated by means of arthroscopic surgery. | 1 year

SECONDARY OUTCOMES:
Determine the correlation of functional outcomes over time in subjects with retears compared with subjects who have an intact cuff repair using the Constant Murley Shoulder Score as well as strength and range of motion. | 1 year
Determination of the correlation between imaging biomarkers (muscle atrophy and fatty infiltration) and the subjects outcome (retear and function). | 1 year
Estimation of the relationship between patient reported outcomes and subject's surgical and functional outcomes. | 1 year
Evaluation of the ability to define | 1 year
Observation of any comorbidity associated with the arthroscopic surgical procedure through the collection of adverse events to provide and SOC reference for future safety studies. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (31):
- United States (31):
  - The Core Institute, Phoenix, Arizona
  - Desert Valley Radiology, Phoenix, Arizona
  - Paradise Valley Hospital, Phoenix, Arizona
  - Banner Boswell Imaging Center, Sun City, Arizona
  - Banner Boswell Medical Center, Sun City, Arizona
  - The Core Institute, Sun City, Arizona
  - Banner Del E Webb Medical Center, Sun City West, Arizona
  - Banner Del E Webb Outpatient Diagnostics, Sun City West, Arizona
  - The CORE Institute-Sun City West, Sun City West, Arizona
  - University of California, San Francisco, San Francisco, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Waltham, Massachusetts
  - Hospital for Special Surgery, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University Orthopaedic Associates, Rochester, New York
  - Cleveland Clinic, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - University Orthopedics, Providence, Rhode Island
  - University Orthopedics, Inc., Providence, Rhode Island
  - Texas Orthopedic Specialists, PA, Bedford, Texas
  - Orthopedic Specialists, Grapevine, Texas
  - Preferred Imaging, Grapevine, Texas
  - Kelsey Research Foundation, Houston, Texas
  - Kelsey-Seybold Spring Medical and Diagnostic Center, Houston, Texas
  - Kelsey Seybold Clinic, Houston, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
  - Harris Methodist Southlake, Southlake, Texas
  - The Everett Clinic, Everett, Washington

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3202V1-1000&StudyName=Arthroscopic%20Surgical%20Outcome%20Study%20In%20Subjects%20With%20Rotator%20Cuff%20Tears